CLINICAL TRIAL: NCT04133974
Title: A Novel Methadone-induced Memory Retrieval-extinction Procedure to Prevent Heroin Craving and Relapse
Brief Title: Methadone Induced Memory Retrieval-extinction Procedure in Heroin Addicts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Dependence, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIDD12035
Record Dates: First submitted 2019-10-14; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Heroin Dependence
MeSH Terms: conditions — Heroin Dependence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Methadone (No Intervention): The subjects take methadone as usual.
- Methadone-10min-Extinction (Experimental): The subjects were given extinction training 10 min following methadone administration.
  Interventions: Behavioral: methadone induced memory retrieval-extinction procedure
- Methadone-6h-Extinction (Sham Comparator): The subjects were given extinction training 6h following methadone administration.
  Interventions: Behavioral: methadone induced memory retrieval-extinction procedure

INTERVENTIONS:
Behavioral: methadone induced memory retrieval-extinction procedure — Drug memory is not invariably stable and can be induced transiently labile again by drug-related cues or drug itself, which is termed as 'reconsolidation'. Previously we and other groups have demonstrated that extinction coincided with reconsolidation weakened the drug memory and decreased drug craving and relapse. In the present study, we tried to interfere the methadone-induced heroin addiction memory reconsolidation by extinction given at different times following methadone administration.
  Arms: Methadone-10min-Extinction; Methadone-6h-Extinction

SUMMARY:
The study assessed the efficacy of a methadone-induced memory retrieval-extinction procedure on heroin craving and relapse. Male participants aged 18-55 years old and prescribed MMT to treat heroin dependence were included in the present study, and randomly assigned to receive methadone, or receive methadone plus 10 minutes plus extinction, or receive methadone plus 6 hours plus extinction. The intervention persisted 3 times per week for 4 weeks. Then the subjects were followed up once a month for cue induced heroin craving and relapse.

DETAILED DESCRIPTION:
In the present study, we explored the effect retrieval-extinction procedure on heroin craving and relapse in heroin addicts using the methadone (a commonly used µ-opioid receptor agonist) instead of heroin as the trigger to reactivate drug memories. The subjects were randomly divided into 3 groups, in which they received methadone alone or extinction sessions 10 min or 6 hours after methadone administration. The extinction sessions were given 3 times per week for 4 weeks, each lasted for 30 min. During the extinction procedure, the subjects were exposed to images, heroin paraphernalia and mimic heroin. Subjective craving, morphine urine test and physiological responses were recorded monthly for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* met the diagnostic criteria of heroin dependence according to DSM-IV
* were prescribed methadone maintenance treatment (MMT) and took it regularly
* no change in city of residence for at least 1 year
* had normal blood pressure and heart rate
* had negative urine morphine screening test
* primary-school level education
* provide signed consent

Exclusion Criteria:

* other substance abuse(except nicotine)
* had a current or past history of Diagnostic and Statistical Manual of Mental Disorders, 4th Edition（DSM-IV) AxisⅠdisorders
* had clinically evident physical disorders
* neurological signs and/or history of neurological disease
* noncompliance with the procedure

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2017-04-23 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
change of cue induced heroin craving | Baseline (Day 0 ), post-intervention (1 month), monthly during follow-up for 4 months (2, 3, 4 and 5 month)
  Heroin craving will be assessed using a visual analog scale (VAS), i.e., an undivided line marked at the left and right ends with 0 ("not at all") and 10 ("extremely high").
change of negative urinary morphine test | Baseline (Day 0), weekly during intervention(1, 2, 3 and 4 week) and monthly during follow-up for 4 months (2, 3, 4 and 5 month)
  All the participants will be required to have urine tests for morphine during screening, weekly during intervention and monthly during follow-up.

SECONDARY OUTCOMES:
cue induced heart rate change | Baseline (Day 0 ), post-intervention (1 month), monthly during follow-up for 4 months (2, 3, 4 and 5 month)
  Heart rate will be monitored immediately before and after cue exposure
cue induced blood pressure change | Baseline (Day 0 ), post-intervention (1 month), monthly during follow-up for 4 months (2, 3, 4 and 5 month)
  Blood pressure will be monitored immediately before and after cue exposure.

IPD SHARING:
Plan to Share IPD: No